CLINICAL TRIAL: NCT01723943
Title: Psychoeducation for Spouses/Partners of Women With Breast Cancer
Brief Title: Educational Counseling in Improving Communication and Quality of Life in Spouses and Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 8061; NCI-2013-01838 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 34500; 8061 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH); R01CA114561 (NIH); NCT02032992 (obsolete NCT alias)
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Anxiety Disorder; Depression; Ductal Breast Carcinoma in Situ; Lobular Breast Carcinoma in Situ; Psychosocial Effects of Cancer and Its Treatment; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage II Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Anxiety Disorders; Depression; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Breast Neoplasms | interventions — Early Intervention, Educational; Methods; Counseling; Psychiatric Rehabilitation; Caregivers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (educational booklet) (Active Comparator): Participants receive the "What's Happening to the Woman I Love?" booklet, which focuses on ways to understand and deal with marital communication and relationship issues arising from breast cancer diagnosis.
  Interventions: Other: educational intervention
- Arm II (Helping Her Heal program) (Experimental): Participants undergo the Helping Her Heal educational counseling program comprising 5 1-hour sessions 2 weeks apart.
  SESSION I: Participants learn stress management skills and discover ways stress affects themselves and their partner.
  SESSION II: Participants practice attentive listening and reduce the tendency to try to distract patients from talking about sad or difficult aspects of the cancer experience.
  SESSION III: Patients learn to help their spouse talk when she is quiet or withdrawn, to add to their understanding of what she is thinking and feeling, and to add to their ways of supporting her during especially difficult times with the cancer.
  SESSION IV: Participants learn strategies for physically reconnecting with spouses.
  SESSION V: Participants review skills from prior sessions, identify strategies he or she will continue to use to manage their personal stress, and identify ways to maintain connection and support.
  Interventions: Other: counseling intervention; Other: educational intervention; Other: psychosocial support for caregiver

INTERVENTIONS:
Other: educational intervention — Receive the "What's Happening to the Woman I Love?" booklet
  Other Names: intervention, educational
  Arms: Arm I (educational booklet)
Other: counseling intervention — Undergo Helping Her Heal educational counseling program
  Other Names: counseling and communications studies
  Arms: Arm II (Helping Her Heal program)
Other: educational intervention — Undergo Helping Her Heal educational counseling program
  Other Names: intervention, educational
  Arms: Arm II (Helping Her Heal program)
Other: psychosocial support for caregiver — Undergo Helping Her Heal educational counseling program
  Arms: Arm II (Helping Her Heal program)

SUMMARY:
This randomized clinical trial studies educational counseling in improving communication and quality of life in spouses and breast cancer patients. An outpatient education and behavior skills training program may help spouses and patients with breast cancer communicate better and improve quality of life. It is not yet known whether educational counseling is more effective than an educational booklet in improving communication and quality of life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test whether the intervention has a beneficial effect on spouses' outcome variables.

II. To test whether the intervention has a beneficial effect on ill partners (patients') outcome variables.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Participants receive the "What's Happening to the Woman I Love?" booklet, which focuses on ways to understand and deal with marital communication and relationship issues arising from breast cancer diagnosis.

ARM II: Participants undergo the Helping Her Heal educational counseling program comprising 5 1-hour sessions 2 weeks apart.

SESSION I: Participants learn stress management skills and discover ways stress affects themselves and their partner.

SESSION II: Participants practice attentive listening and reduce the tendency to try to distract patients from talking about sad or difficult aspects of the cancer experience.

SESSION III: Patients learn to help their spouse talk when she is quiet or withdrawn, to add to their understanding of what she is thinking and feeling, and to add to their ways of supporting her during especially difficult times with the cancer.

SESSION IV: Participants learn strategies for physically reconnecting with spouses.

SESSION V: Participants review skills from prior sessions, identify strategies he or she will continue to use to manage their personal stress, and identify ways to maintain connection and support.

After completion of study, patients are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Spouses (in both heterosexual couples and same-sex couples) of women diagnosed within the past 6 months with stage 0, I, II or III breast cancer (in situ/local/regional disease) will be eligible to participate, as will the diagnosed wife/partner
* Spouses and patients must be married or cohabiting for at least 6 months
* Spouses and patients must have English as one of their languages of choice (they can be multilingual)
* Spouses and patients must live within 25 miles of the University of Washington (UW) study center
* Spouses/partners must be willing to give a sample of blood and/or sputum at time of first and second data collections

Exclusion Criteria:

* Woman diagnosed with stage IV or recurrent breast cancer or who is > 6 months post-diagnosis
* Woman and/or spouse not able to read and write in English
* Spouses could not participate if the ill partner refused participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2009-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in State-Trait Anxiety Inventory (STAI) spouse scores | Baseline to 8 weeks
  The primary analysis will be multivariate analysis of covariance (MANCOVA) with 3 outcome variables, controlling for baseline values and additional covariates identified during the preparatory analyses. Further analyses done on each outcome variable separately to determine if the outcome had a stronger effect on some. Secondary analyses will include analysis of covariance (ANCOVA).
Change in Center for Epidemiologic Studies Depression Scale (CES-D) spouse scores | Baseline to 8 weeks
  The primary analysis will be MANCOVA with 3 outcome variables, controlling for baseline values and additional covariates identified during the preparatory analyses. Further analyses done on each outcome variable separately to determine if the outcome had a stronger effect on some. Secondary analyses will include ANCOVA.
Change in STAI patient scores | Baseline to 8 weeks
  The primary analysis will be MANCOVA with 3 outcome variables, controlling for baseline values and additional covariates identified during the preparatory analyses. Further analyses done on each outcome variable separately to determine if the outcome had a stronger effect on some. Secondary analyses will include ANCOVA.
Change in CES-D patient scores | Baseline to 8 weeks
  The primary analysis will be MANCOVA with 3 outcome variables, controlling for baseline values and additional covariates identified during the preparatory analyses. Further analyses done on each outcome variable separately to determine if the outcome had a stronger effect on some. Secondary analyses will include ANCOVA.

SECONDARY OUTCOMES:
Change in spouse/partner Skills Checklist scores | Baseline to 8 weeks
  Secondary analyses will use ANCOVA, controlling for baseline variables, to test for intervention versus control differences. A significant improvement in an intermediate outcome variable would be consistent with that variable being a mediator of the treatment effect on the primary outcomes.
Change in spouse/partner CASE scores | Baseline to 8 weeks
  Secondary analyses will use ANCOVA, controlling for baseline variables, to test for intervention versus control differences. A significant improvement in an intermediate outcome variable would be consistent with that variable being a mediator of the treatment effect on the primary outcomes.
Change in spouse/partner Mutuality and Interpersonal Sensitivity Scale (MIS) scores | Baseline to 8 weeks
  Secondary analyses will use ANCOVA, controlling for baseline variables, to test for intervention versus control differences. A significant improvement in an intermediate outcome variable would be consistent with that variable being a mediator of the treatment effect on the primary outcomes.
Change in patient MIS scores | Baseline to 8 weeks
  Secondary analyses will use ANCOVA, controlling for baseline variables, to test for intervention versus control differences. A significant improvement in an intermediate outcome variable would be consistent with that variable being a mediator of the treatment effect on the primary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Lewis, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Lewis FM, Griffith KA, Alzawad Z, Dawson PL, Zahlis EH, Shands ME. Helping Her Heal: Randomized clinical trial to enhance dyadic outcomes in couples. Psychooncology. 2019 Feb;28(2):430-438. doi: 10.1002/pon.4966. Epub 2018 Dec 28. PMID 30549145